CLINICAL TRIAL: NCT00246129
Title: A Randomised Controlled Comparison of Campath-Tacrolimus vs IL2R MoAb-Tacrolimus/Mycophenolate Mofetil in Kidney Transplantation
Brief Title: CamTac Trial:Campath-Tacrolimus vs IL2R MoAb/Tacrolimus/MMF in Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMagnusson (Other)
Responsible Party: Sponsor-Investigator, EMagnusson, RIO, Imperial College Healthcare NHS Trust
Organization: Imperial College Healthcare NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMHREN0501; 2005-002856-17 (EudraCT Number)
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Kidney Transplantation; Kidney Diseases; Kidney Failure
Keywords: Kidney Transplantation; Kidney Disease; Kidney Failure; Graft Rejection
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency | interventions — Alemtuzumab; Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Campath-Tacrolimus (Active Comparator): Campath induction with 7-day short-course steroids followed by tacrolimus monotherapy
  Interventions: Drug: Campath
- Daclizumab-Tacrolimus-Mycophenolate (Experimental): Daclizumab induction with 7-day short-course steroids followed by Tacrolimus and Mycophenolate mofetil therapy
  Interventions: Drug: Daclizumab

INTERVENTIONS:
Drug: Campath — Monoclonal antibody induction therapy
  Other Names: Alemtuzumab
  Arms: Campath-Tacrolimus
Drug: Daclizumab — Monoclonal antibody induction therapy
  Other Names: Zinbryta
  Arms: Daclizumab-Tacrolimus-Mycophenolate

SUMMARY:
The advent of new, potent immunosuppressive (anti-rejection) drugs over the past ten years has substantially reduced the risk of rejection after kidney transplantation, has allowed the development of immuno-suppressive regimens that do not use long-term steroids (steroid avoidance), and has improved transplant success rates both in the short and medium term.

The main new agents used in these modern regimens are the calcineurin inhibitor (CNI) tacrolimus; the anti-proliferative agent mycophenolate; and induction agents which are used to provide effective early suppression of the rejection process; these include monoclonal antibodies (MoAb) such as IL-2 receptor blocking antibodies (IL-2R MoAb: basiliximab and daclizumab) and the anti-CD52 antibody Campath-1H (alemtuzumab).

Although almost all modern immunosuppressive regimens involve one or more of these agents, it is not known which is the safest and most effective combination.

This randomised controlled trial compares two steroid sparing regimens which have been used with very good short and medium term results at St Mary's Hospital Renal and Transplant Unit over the last 5 years. The primary hypothesis is that the alemtuzumab/tacrolimus regimen is as effective and safe as the IL-2R MoAb/tacrolimus/mycophenolate regimen.

DETAILED DESCRIPTION:
RECENT EXPERIENCE AT ST MARY'S:

The St Mary's Hospital Renal Unit (now combined with the Hammersmith Hospital Renal Unit at the West London Renal and Transplant Centre) introduced Tacrolimus based immunosuppression in 1995, developing a steroid avoidance regimen based on Tacrolimus, Mycophenolate, and IL-2R MoAb between 2000 and 2002, and moving to Campath-1H as an induction agent in 2004. Results over this period have been excellent with five and ten year survivals with functioning graft rates of 82% and 72% for the first 260 cadaveric kidney transplants performed since 1995.

The two most recent regimens used at St Mary's have both produced very low (< 10%) rejection rates, and very good (> 90%) short-term rejection-free patient and graft survival rates. Between 2002 and 2004, the regimen consisted of induction with an Interleukin-2 (IL2) -Receptor blocking monoclonal antibody with Tacrolimus and Mycophenolate as long term maintenance therapy. In patients without rejection steroid usage was limited to the first 7 days post-transplant. The current regimen uses Campath-1H (which is now well established as an induction agent in renal transplantation for induction), with Tacrolimus monotherapy maintenance and an identical short-course steroid regimen.

CHARACTERISTICS OF THE TWO REGIMENS TO BE COMPARED:

The IL2R MoAb/Tacrolimus/Mycophenolate/Short-course steroids regimen (2002-2004 Regimen 1) has the advantage of flexibility in terms of adjusting maintenance therapy to allow clinical response to patients and transplants with different tolerance of the two maintenance agents, but involves increased expense in terms of using and monitoring the blood levels of two modern (and hence expensive) agents. In addition, patients have long-term exposure to the anti-proliferative agent Mycophenolate, which can be associated with increased risk of infection, gastrointestinal side effects, and skin malignancies.

The Campath-1H/Tacrolimus/Short-course steroids regimen (2004-current, Regimen 2) has the advantage of highly effective immunosuppression in the initial 3-month period, allowing lower doses of the potentially nephrotoxic Tacrolimus to be used, and simplicity, but exposes patients to a period of several months of lymphopenia (reduced lymphocyte counts in the blood) after Campath administration, and reliance on Tacrolimus monotherapy for maintenance which might lead to greater long term Tacrolimus exposure.

PROPOSED STUDY:

In order to allow a proper comparison of these two anti-rejection treatment combinations we propose a randomised trial which will enable us to consider the relative merits of the two regimens without the introduction of bias associated with using historical control groups. Transplant recipients will be randomised in a 1:2 ratio to regimen 1 and regimen 2.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients under the care of the West London Renal and Transplant Centre

Exclusion Criteria:

* Patients who are unable to give written informed consent
* Simultaneous kidney/pancreas transplant recipients
* Non-heart beating deceased donor transplant recipients
* Patients who would not be offered Campath-1H induction under our current protocol (patients with previous malignancy or with previous exposure to cytotoxic or antiproliferative agents)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2005-10 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam G McLean, FRCP, DPhil, Principal Investigator — Hammersmith Hospital NHS Trust; David H Taube, MBBCh, FRCP, Study Director — Hammersmith Hospital NHS Trust
Locations (1):
- West London Renal and Transplant Centre, 4th Floor Ham House, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loucaidou M, McLean AG, Cairns TD, Griffith M, Hakim N, Palmer A, Papalois V, Van Tromp J, Loucaides C, Welsh KI, Taube D. Five-year results of kidney transplantation under tacrolimus-based regimes: the persisting significance of vascular rejection. Transplantation. 2003 Oct 15;76(7):1120-3. doi: 10.1097/01.TP.0000076474.76480.A4. PMID 14557763
- [Background] Borrows R, Loucaidou M, Van Tromp J, Cairns T, Griffith M, Hakim N, McLean A, Palmer A, Papalois V, Taube D. Steroid sparing with tacrolimus and mycophenolate mofetil in renal transplantation. Am J Transplant. 2004 Nov;4(11):1845-51. doi: 10.1111/j.1600-6143.2004.00583.x. PMID 15476485
- [Background] Borrows R, Loucaidou M, Van Tromp J, Singh S, Cairns T, Griffith M, Hakim N, McLean A, Palmer A, Papalois V, Taube D. Steroid sparing in renal transplantation with tacrolimus and mycophenolate mofetil: three-year results. Transplant Proc. 2005 May;37(4):1792-4. doi: 10.1016/j.transproceed.2005.03.150. PMID 15919468
- [Result] Chan K, Taube D, Roufosse C, Cook T, Brookes P, Goodall D, Galliford J, Cairns T, Dorling A, Duncan N, Hakim N, Palmer A, Papalois V, Warrens AN, Willicombe M, McLean AG. Kidney transplantation with minimized maintenance: alemtuzumab induction with tacrolimus monotherapy--an open label, randomized trial. Transplantation. 2011 Oct 15;92(7):774-80. doi: 10.1097/TP.0b013e31822ca7ca. PMID 21836540

RESULTS

PARTICIPANT FLOW:
Groups:
- Campath-Tacrolimus: Campath (1x30mg) induction with 7-day short-course steroids followed by tacrolimus monotherapy (dose adjusted to target trough level 9-11ng/ml)
- Daclizumab-Tacrolimus-Mycophenolate: Daclizumab 2mg/kg x2 days 0+14) induction with 7-day short-course steroids followed by Tacrolimus (adjusted to target trough 9-11ng/ml) and Mycophenolate mofetil therapy (750mg bd)
Period: Overall Study
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Started | 82 | 41
Completed | 75 | 39
Not Completed | 7 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 2 | 1
Not completed — suffered primary non-function | 1 | 0
Not completed — grafts failed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate | Total
Number analyzed (Participants) | 82 | 41 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 39 | 116
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (13.4) | 47.0 (10.6) | 47.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 14 | 42
  Male | 54 | 27 | 81
Region of Enrollment [Number; unit: participants]
  United Kingdom | 82 | 41 | 123

OUTCOME MEASURES:

1. Primary Outcome: One Year Survival With a Functioning Graft
Description: One year survival with a functioning graft, defined as transplant recipient remaining alive and dialysis-independent. the functioning graft is a graft still functioning at the time of analysis.
  Graft function was estimated using the Modification of Diet in Renal Disease four-variable formula and comparison of graft function between arms undertaken with Student'st test.
Time Frame: 1 year
Measure: Number (90% Confidence Interval); unit: Percent of patients
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 82 | 41
Percent of patients | 97.6 [90.6 to 99.4] | 95.1 [81.9 to 98.8]
Statistical Analysis 1: Comparison: Campath-Tacrolimus vs Daclizumab-Tacrolimus-Mycophenolate; Test type: Superiority; p = 0.467, Log Rank

2. Secondary Outcome: Occurrence of Rejection Episodes
Description: Biopsy-proven rejection episodes classified using Banff criteria
Time Frame: 1 year
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Groups:
- Campath Tacrolimus: Alemtuzumab induction with short-course steroids and Tacrolimus maintenance monotherapy
Arm/Group | Campath Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 82 | 41
Percentage of patients | 91.2 [82.4 to 95.7] | 82.3 [66.4 to 91.1]
Statistical Analysis 1: Comparison: Campath Tacrolimus vs Daclizumab-Tacrolimus-Mycophenolate; Test type: Superiority; p = 0.138, Log Rank

3. Secondary Outcome: Occurrence of Significant Episodes of Infection
Description: Occurence of infection of sufficient severity to produce positive cultures or Nucleic-acid test results from blood, urine, or other body fluids
Time Frame: 1 year
Measure: Number; unit: # of occurrences per 100 patient years
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 82 | 41
# of occurrences per 100 patient years | 73 | 76

4. Secondary Outcome: Initial Length of Stay in Hospital
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 82 | 41
Days | 11.7 (6.4) | 12.1 (7.6)

5. Secondary Outcome: Presence in the Blood of Cells Which Might Trigger Rejection in, or Promote Tolerance to the Graft
Time Frame: 3 years
Population: Data not collected
Arm/Group | Campath Tacrolimus ' | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Early Development of Scarring in the Grafts
Description: Biopsy proven Calcineurin Inhibitor (CNI) toxicity free survival
Time Frame: 1 year
Measure: Number; unit: Percentage of participants with no scar
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 82 | 41
Percentage of participants with no scar | 96 | 90

7. Secondary Outcome: Graft Function: Level of Creatinine
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 82 | 41
mmol/L | 127.3 (36.2) | 147.0 (69.1)

8. Secondary Outcome: Patient Survival Censored for Death With Function
Description: Cumulative patient survival
Time Frame: 2 years
Measure: Number; unit: Percentage of transplant recipients
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 82 | 41
Percentage of transplant recipients | 98 | 98

9. Secondary Outcome: Graft Survival Censored for Death With Function
Description: Graft survival (defined as grafts maintaining dialysis independence)
Time Frame: 2 years
Measure: Number; unit: Percentage of grafts
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
Number analyzed (Participants) | 82 | 41
Percentage of grafts | 91 | 95

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Campath-Tacrolimus | Daclizumab-Tacrolimus-Mycophenolate
All-Cause Mortality (participants affected / at risk) | 2/82 | 1/41
Serious Adverse Events (participants affected / at risk) | 5/82 | 5/41
Other Adverse Events (participants affected / at risk) | 59/82 | 30/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath-Tacrolimus (N=82) | Daclizumab-Tacrolimus-Mycophenolate (N=41)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — ITP
New-onset diabetes after transplantation (Metabolism and nutrition disorders) | 4 (4) | 5 (5) — NODAT
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath-Tacrolimus (N=82) | Daclizumab-Tacrolimus-Mycophenolate (N=41)
Urinary tract infection (Infections and infestations) | 31 (31) | 9 (9)
Bacteremia (Infections and infestations) | 15 (15) | 9 (9)
Wound infection (Infections and infestations) | 6 (6) | 6 (6)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 4 (4)
Other infection (Infections and infestations) | 6 (6) | 2 (2)

LIMITATIONS AND CAVEATS:
Our trial was conservatively powered to detect a large difference in survival with a functioning graft at 1 year, so we are not able to exclude the possibility of small differences, the single-centre nature of the study may limit it's applicability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No